CLINICAL TRIAL: NCT01749852
Title: Effect of Polyphenol-rich Dark Chocolate on Body Weight in Overweight and Obese Adults: A Pilot Study
Brief Title: Effect of Polyphenol-rich Dark Chocolate on Body Weight in Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Margaret University (Other)
Collaborators: Barry Callebaut (Unknown)
Responsible Party: Principal Investigator, Grace Farhat, PhD research student, Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DC-BW 01
Record Dates: First submitted 2012-12-10; First posted 2012-12-17 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2013-05

CONDITIONS: Body Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyphenol-rich Dark chocolate (Experimental): Dark chocolate with 500 mg of polyphenols
  Interventions: Other: Polyphenol-rich Dark chocolate
- Placebo Dark chocolate (Placebo Comparator): This chocolate contains little or no polyphenols
  Interventions: Other: Placebo Dark chocolate

INTERVENTIONS:
Other: Polyphenol-rich Dark chocolate — Participants will be asked to consume 20g of dark chocolate containing 500mg of polyphenols daily for a period of 12 weeks
  Arms: Polyphenol-rich Dark chocolate
Other: Placebo Dark chocolate — Participants will be asked to consume 20g of dark chocolate containing little or no polyphenols for a period of 12 weeks
  Arms: Placebo Dark chocolate

SUMMARY:
The aim of this study is to investigate if dark chocolate rich in polyphenols decreases body weight/ body fat in the overweight and obese adult population.

DETAILED DESCRIPTION:
Polyphenols are phytochemicals widely available in plants, and may have several favourable effects on health. Dark chocolate (DC) is one of the highest sources of polyphenols in foods. Animal and in vitro studies have demonstrated that cocoa and dark chocolate may exert anti-obesity effects mainly due to the polyphenol effect on glucose and fatty acid metabolism. Human studies have showed that regular chocolate eaters have a lower body weight compared to non regular eaters, and that DC promotes satiety and reduces cravings. The aim of this pilot study is to investigate the effect of polyphenol-rich DC on body weight in the overweight and obese adult population, when incorporated into a non-restricted diet. Twenty-eight apparently healthy volunteers will be recruited. Participants will randomly receive 20g daily of one of the two different types of DC: Placebo DC (low in polyphenols) or DC rich in polyphenols (500mg) for a period of twelve weeks. Participants will be asked to make three appointments and one follow-up appointment to the university clinical lab. Anthropometric measurements (height, weight, waist circumference, body fat percentage) will be taken during each visit. Compliance will be defined by the intake of 85 % or more of the chocolate weekly, and will be tested by the measure of total polyphenols in a 24-hour urine sample before, during and at the end of the intervention. To monitor any fluctuations in the participants' diet or physical activity during the study period, a three-day diet diary, a Food Frequency questionnaire assessment for polyphenol intake and a physical activity questionnaire will be collected before the start of the study and every four weeks. A follow-up appointment (four weeks after the end of intervention) will check if any differences in anthropometric measures have been maintained. Data will be analysed with an ANCOVA with time (pre- and post-) and treatment (DC and placebo) as between-subject factor. This study will have novel findings and will be the basis for a future larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* BMI between 25-35
* Males and Females
* Age: 18-65 years

Exclusion Criteria:

* Participants with cardiovascular diseases, hypertension or diabetes
* Participants taking any medications that affect insulin, cholesterol, triglycerides or Blood pressure
* Participants who recently participated or are currently on a weight management program
* Participants with regular consumption of cocoa or DC (> 1 serving/week)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in Body weight | Baseline, week 6, week 12 and week 16
  The body weight will be measured using a digital scale

SECONDARY OUTCOMES:
Change in Body Fat percentage | Baseline, week 6, week 12 and week 16
Change in Waist circumference | Baseline, week 6, week 12 and week 16
Change in urinary Cortisol-to-cortisone ratio | Baseline, week 6 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Emad Al-Dujaili, PhD, Study Director — Queen Margaret University
Locations (1):
- Queen Margaret University Lab, Musselburgh, East Lothian, United Kingdom